CLINICAL TRIAL: NCT04805567
Title: Adenoma Miss Rate in Tandem Endocuff-assisted Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Venizelio General Hospital (Other)
Responsible Party: Principal Investigator, Maria Fragaki, MD, PhD, Venizelio General Hospital
Other Study IDs: VenizelioGH
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Colon Polyp; Endocuff
Keywords: endocuff; tandem colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with polyps and adenomas: The inclusion criteria are: (i) CRC screening; (ii) post-polypectomy surveillance; (iii) diagnostic assessment (anemia, lower gastrointestinal bleeding, abdominal pain, recent change in bowel habits); and (iv) age over 50 years.
  Interventions: Device: endocuff

INTERVENTIONS:
Device: endocuff — The Endocuff is a device that can be mounted on the tip of an endoscope and may assist to inspect a greater surface of the colonic mucosa by pulling backwards, flattening, and stretching the colonic folds as the endoscope is gradually withdrawn.

SUMMARY:
Colonoscopy is a valuable tool in reducing the incidence and mortality from colorectal cancer (CRC). Older back-to-back studies evaluating novel endoscopes indicated that conventional colonoscopy misses almost 20% of adenomas. In order to improve the diagnostic accuracy of colonoscopy and to improve the adenoma detection rate (ADR) (a significant marker of quality), efforts have been made to improve endoscopic techniques, the bowel preparation, to keep slower withdrawal time, and to use new technologies and devices. Since 2012, a new accessory device (Endocuff; ARC Medical Design, Leeds, UK), which is mounted on the tip of the colonoscope has been introduced to the market. The Endocuff is a device that can be mounted on the tip of an endoscope and may assist to inspect a greater surface of the colonic mucosa by pulling backwards, flattening, and stretching the colonic folds as the endoscope is gradually withdrawn. Use of this device may achieve better visualization of the bowel lumen, especially behind folds, and improve stability of the instrument on withdrawal.

The aim of this study is to conduct a back-to-back endoscopy study and to evaluate the contribution of Endocuff-assisted colonoscopy to the detection of missed adenomas in a mixed population of colorectal cancer (CRC) screening/surveillance and symptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* (i) CRC screening; (ii) post-polypectomy surveillance; (iii) diagnostic assessment (anemia, lower gastrointestinal bleeding, abdominal pain, recent change in bowel habits); and (iv) age over 50 years.

Exclusion Criteria:

* (i) age below 50 years; (ii) the presence of significant comorbidities (American Society of Anesthesiologists [ASA] score III or IV); (iv) recent abdominal surgery; (iv) inflammatory bowel disease; (v) colectomy; (vi) polyposis syndrome; (vii) the presence of acute, severe colitis or a known colonic stricture (viii) boston scale bowel preparation ≥6.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Τhe study is a single center cohort study. Venizeleio General Hospital is a tertiary hospital and the population that will be selected would be residents of the island of Crete.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
of Endocuff-assisted colonoscopy adenoma and polyp miss rate | up to 21 days after the colonoscopy
  The primary outcome is the measurement of Endocuff-assisted colonoscopy adenoma and polyp miss rates, overall and in the proximal colon.

IPD SHARING:
Plan to Share IPD: No